CLINICAL TRIAL: NCT00858949
Title: Time-Motion Study of PONV Costs in Ambulatory Surgery
Brief Title: Costs of Postoperative Nausea and Vomiting in Ambulatory Surgery Patients
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 08-415
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Outpatient surgery; Postoperative nausea and vomiting; Costs; Observational
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post surgery monitored group: Outpatients undergoing elective surgery with anesthesia that is expected to last one hour and to require significant postoperative opioids

SUMMARY:
This is an observational study with the goal of determining the costs of nausea and vomiting in ambulatory patients after surgery from the US societal perspective.

DETAILED DESCRIPTION:
The direct cost between the end of outpatient surgery and discharge from the hospital will include costs of labors and supplies for any outpatient care, physician visits, laboratory tests, and prescribed medications, which may be used to treat operation side effects. Based on the time and motion study design, the timing of these healthcare activities will be collected. The study coordinator will observe the actual time taken for each activity for each patient. The observation period will begin after completion of the outpatient surgery. The start and end times for each activity performed will be recorded. Therefore, each activity and its duration will be concurrently recorded. We will also query patients daily to determine additional costs associated with PONV until the third postoperative morning.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* American Society of Anesthesiologists (ASA) physical status 1 to 3
* Outpatients undergoing elective surgery with anesthesia that is expected to last one hour and to require significant postoperative opioids
* Patients must provide written informed consent and have at least two of the following PONV risk factors: (1) female gender, (2) history of PONV and/or currently prone to motion sickness, (3) non smoking status.

Exclusion Criteria:

* Any drug with potential antiemetic efficacy within 24 hours prior to the anesthetic procedure
* Vomiting, retching, or nausea in the 24 hours preceding anesthesia
* Body mass index >40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients undergoing elective surgery with anesthesia that is expected to last one hour and to require significant postoperative opioids
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the costs of PONV in ambulatory patients from the US societal perspective | 72 hours post op

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States